CLINICAL TRIAL: NCT05179733
Title: The Efficacy and Safety of Zanubrutinib, Rituximab and Lenalidomide (ZR2) Versus Rituximab Combined With Low-dose CHOP (R-miniCHOP) in the Treatment of Unfit or Frail de Novo Diffuse Large B-cell Lymphoma Patients Aged Older Than or Equal to 70 Years: A Multicenter, Prospective, Randomized, Open-label, Controlled Trial
Brief Title: The Efficacy and Safety of ZR2 Versus R-miniCHOP in the Treatment of Unfit or Frail de Novo Diffuse Large B-cell Lymphoma Patients Aged Older Than or Equal to 70 Years
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Ningbo No. 1 Hospital (Other); National Naval Medical Center (U.S. Federal Agency); Shanghai Fengxian District Central Hospital (Other); YANCHENG NO.1 PEOPLE'S HOSPITAL (Unknown); The First Affiliated Hospital of Nanchang University (Other); Affiliated Hospital of Nantong University (Other); Sir Run Run Shaw Hospital (Other); Northern Jiangsu People's Hospital (Other); The First People's Hospital of Changde City (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Changzhou No.2 People's Hospital (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Huai'an First People's Hospital (Other); Taizhou Hospital (Other); The First People's Hospital of Kunshan (Other); First Affiliated Hospital of Fujian Medical University (Other); Huadong Hospital (Other); Henan Provincial People's Hospital (Other); First Hospital of China Medical University (Other); Shandong Provincial Hospital (Other Government); HARBIN THE FIRST HOSPITAL (Unknown); The First Hospital of Jilin University (Other); Hunan Cancer Hospital (Other); Qilu Hospital of Shandong University (Other); THE FIRST AFFILIATED HOSPITAL (Unknown); The Second Affiliated Hospital of Dalian Medical University (Other); SUZHOU HONGCI HEMATOLOGY HOSPITAL (Unknown)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director, Hematology Department, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHL-014
Record Dates: First submitted 2021-11-22; First posted 2022-01-05 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Diffuse Large B-Cell Lymphoma; Elderly patients; Zanubrutinib; Lenalidomide; Rituximab; R-miniCHOP
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ZR2 (Experimental): six courses of zanubrutinib, rituximab and lenalidomide
  Interventions: Drug: six courses of zanubrutinib, rituximab and lenalidomide
- R-miniCHOP (Active Comparator): six courses of rituximab combined with low-dose CHOP
  Interventions: Drug: six courses of rituximab combined with low-dose CHOP

INTERVENTIONS:
Drug: six courses of zanubrutinib, rituximab and lenalidomide — Patients in ZR2 group will receive 6 cycles of zanubrutinib 160mg bid, day 1-21, orally, lenalidomide 25mg qd, day 2-11, orally, rituximab 375mg/m², day 1, intravenously, every 21 days.
  Arms: ZR2
Drug: six courses of rituximab combined with low-dose CHOP — Patients in R-miniCHOP group will receive rituximab 375 mg/m² on day 1, cyclophosphamide 400 mg/m², doxorubicin 25 mg/m², and vincristine 1 mg on day 2, and prednisone 40 mg/m² on days 2-6, every 21 days.
  Arms: R-miniCHOP

SUMMARY:
A multicenter, prospective, randomized, open-label, controlled trial to evaluate the efficacy and safety of zanubrutinib, rituximab and lenalidomide (ZR2) versus rituximab combined with low-dose CHOP (R-miniCHOP) in the treatment of unfit or frail de novo diffuse large B-cell lymphoma patients aged older than or equal to 70 years

DETAILED DESCRIPTION:
This study will evaluate the efficacy and safety of ZR2 versus R-miniCHOP in the treatment of unfit or frail de novo diffuse large B-cell lymphoma patients aged older than or equal to 70 years. Subjects will be randomly assigned 1:1 to ZR2 or R-miniCHOP regimen. The stratification will be performed according to international prognostic index (0-2 / 3-5).

Patients in ZR2 group will receive 6 cycles of zanubrutinib 160mg bid, day 1-21, orally, lenalidomide 25mg qd, day 2-11, orally, rituximab 375mg/m², day 1, intravenously, every 21 days. Patients in R-miniCHOP group will receive rituximab 375 mg/m² on day 1, cyclophosphamide 400 mg/m², doxorubicin 25 mg/m², and vincristine 1 mg on day 2, and prednisone 40 mg/m² on days 2-6, every 21 days.

ELIGIBILITY:
Inclusion Criteria

Patients must satisfy all of the following criteria to be enrolled in the study:

* Histologically-confirmed diffuse large B-cell lymphoma (without central nervous system involvement)
* Eastern Cooperative Oncology Group performance status 0-3
* Aged ≥ 80 years old or aged 70-79 with comprehensive geriatric assessment stratified as unfit or frail
* International normalized ratio and activated partial thromboplastin time are both 1.5 times lower than the upper limits of normal (ULN).
* At least 1 measurable site of disease (defined as lymph nodes with the long diameters longer than 1.5cm, or extra-nodal sites with the long diameters longer than 1.0cm; meanwhile, any lesion site with at least 2 measurable vertical diameters)
* Life expectancy of at least 3 months determined by researchers
* The patient or his or her legal representative must provide written informed consent prior to any special examination or procedure for the research.
* Anti-lymphoma drugs have not been used before (except glucocorticoids).

Exclusion criteria

Presence of any of the following criteria will exclude a patient from enrollment:

* Uncontrolled cardio- and cerebro-vascular disease, blood clotting disorders, connective tissue diseases, serious infectious diseases and other diseases
* Laboratory measures meet the following criteria at screening (unless caused by lymphoma):

  1. Neutrophils<1.5×10^9/L
  2. Platelets<80×10^9/L (Platelets<50×10^9/L in case of bone marrow involvement)
  3. ALT or AST is 2 times higher than the upper limits of normal (ULN), AKP and bilirubin are 1.5 times higher than the ULN.
  4. Creatinine is 1.5 times higher than the ULN or eGFR is lower than 40ml/min/1.73m^2 (according to Cockcroft-Gault Equation or MDRD Equation).
* HIV-infected patients
* Left ventricular ejection fraction<50%
* Patients with HbsAg positive are required to have HBV DNA<1.0×10^3 IU/ml before entering the group. In addition, if the patient is HBsAg negative but HBcAb positive (regardless of HBsAb status), HBV DNA test is also required, and HBV DNA<1.0×10^3 IU/ml is required before entering the group.
* Other anti-tumor treatments (lymphoma or other types of tumors) are currently in progress.
* Patients with psychiatric disorders or patients who are known or suspected to be unable to fully comply with the study protocol
* Require treatment with strong/moderate CYP3A inhibitors or inducers.
* History of stroke or intracranial hemorrhage within 6 months prior to start of therapy
* Inability to swallow capsules or presence of diseases that significantly affect gastrointestinal function, such as malabsorption syndrome, post-bariatric surgery, inflammatory bowel disease and complete or incomplete intestinal obstruction
* Other medical conditions determined by the researchers that may affect the study

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Baseline up to data cut-off (up to approximately 2 years)
  Progression-free survival was defined as the time from the date of randomization until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Complete response rate | At the end of Cycle 6 (each cycle is 21 days)
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Overall survival | Baseline up to data cut-off (up to approximately 2 years)
  Overall survival was defined as the time from the date of randomization to the date of death from any cause.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From enrollment to study completion, a maximum of 4 years
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Percentage of Participants Achieving Meaningful Improvement in European Organisation for Research and Treatment of Cancer Quality of Life-Core 30 Questionnaire (EORTC QLQ-C30) | Day 1 of Cycles 1 and 4 (Cycle length=21 days); 30 days after treatment completion
  Quality of Life will be assessed by EORTC QLQ-C30 (Verison 3.0).
Percentage of Participants Achieving Meaningful Improvement in EORTC QLQ-ELD14 (Elderly Module) | Day 1 of Cycles 1 and 4 (Cycle length=21 days); 30 days after treatment completion
  Quality of Life will be assessed by EORTC QLQ-ELD14.
Percentage of Participants Achieving Meaningful Improvement in Functional Assessment of Cancer Therapy-Lymphoma Lymphoma Subscale (FACT-Lym LymS) | Day 1 of Cycles 1 and 4 (Cycle length=21 days); 30 days after treatment completion
  Quality of Life will be assessed by FACT-Lym LymS.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No